CLINICAL TRIAL: NCT01024829
Title: Dose Escalation by Boosting Radiation Dose Within the Primary Tumor on the Basis of a Pre-treatment FDG-PET-CT Scan in Stage IB, II and III NSCLC: a Randomized Phase II Trial
Brief Title: Dose Escalation by Boosting Radiation Dose Within the Primary Tumor Using FDG-PET-CT Scan in Stage IB, II and III NSCLC
Acronym: PET Boost
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PET Boost
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: NSCLC
Keywords: Non small cell lung cancer; Inoperable; HX4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole tumor boost (Other): Patients in this arm will receive radiotherapy (66Gy) in 24 fractions of 2.75 Gy with an integrated boost to the primary tumor as a whole
  Interventions: Radiation: Radiotherapy
- Boost 50% SUV area (Other): Patients in this arm receive radiotherapy (66Gy) in 24 fractions of 2.75Gy with an integrated boost to the 50% SUVmax area of the primary tumor (of the pre-treatment FDG-PET-CT scan)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy

SUMMARY:
Increasing ("boosting") the radiation dose for patients with non-small cell lung carcinoma to the individual maximal dose which can safely be given. The question is if patients should receive this boost on the whole tumor on part of the tumor. Therefore patients are randomized for one of these two treatment options. All patients will receive 24 radiations. Dose increasement will be enabled by a so called integrated boost.

Furthermore:

- PET imaging of hypoxia using [18F]HX4, single injection and then PET CT scanning two and four hours post injection.

DETAILED DESCRIPTION:
A randomized phase II study will be conducted in patients with inoperable stage IB, II or III non-small cell lung cancer (NSCLC). The patients will be randomized to receive the standard 66 Gy given in 24 fractions of 2.75 Gy with an integrated boost to the primary tumor as a whole (Arm A) or with an integrated boost to the 50% SUVmax area of the primary tumor (of the pre-treatment FDG-PET scan) (Arm B). Both treatment arms may be combined with chemotherapy (concurrent or sequential). Patients fulfilling the eligibility criteria will be registered in the study, and an initial radiotherapy treatment planning will be performed. When an integrated boost to the primary tumor as a whole up to 72 Gy is not possible because of dose constraints, the patient will receive 66 Gy or lower according to the normal tissue tolerance (see below). They will not be randomized, but will be followed in the trial. As such, it will be clear which proportion of patients can receive an integrated boost and what the outcome is when dose-escalation is not possible.

Stage IB-II patients receive radiotherapy alone, and stage III patients combined chemotherapy and radiation. The patients may have received induction chemotherapy up to two cycles before registration in this trial. The statistical calculations have been performed to deal with this patient heterogeneity.

The primary objective of this study is to determine the local progression-free survival (LPFS)at 1 year.

Secondary objectives will be

* Toxicity as a function of radiotherapy dose and volume of the tissue irradiated.
* Overall survival.
* Quality of life

Furthermore:

* PET imaging of hypoxia using [18F]HX4, single injection and then PET CT scanning two and four hours post injection.
* Dynamic Contrast-Enhanced CT imaging

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years with any subtype of pathologically proven (biopsy or cytology), non-small cell lung cancer. The diagnosis may be established from biopsy or cytology obtained from the primary tumor and/ or from metastatic lymph nodes.
2. Minimal diameter of the primary tumor 4 cm, this to allow for boosting of sub-volumes.
3. UICC TNM Stage T2-4, N0-3, M0 disease (TNM definition see appendix 2).
4. Only stage IB-II patients who are nog candidates for surgery are study candidates.
5. Measurable disease at registration.
6. ECOG-performance status ≤ 2 (see appendix 6)
7. Lung function: FEV1 and DLCO at least 40 % of the age-adjusted normal value
8. Willing and able to give a written informed consent.
9. Patients with locoregional recurrent lung tumor following surgery or a second primary cancer (at least 3 years after treatment) are eligible, unless a pneumonectomy was performed.
10. SUVmax in the pre-treatment FDG-PET scan ≥ 5 for the primary tumor.
11. Adequate organ function, including the following:

    * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, and hemoglobin ≥ 9 g/dL.
    * Hepatic: bilirubin ≤ 1.5 times the upper limit of normal (x ULN); alkaline phosphatase (AP), aspartate aminotransferase (ASAT), and alanine aminotransferase (ALAT) ≤ 3.0 x ULN (AP, AST, and ALT ≤ 5 x ULN is acceptable if liver has tumor involvement).
    * Renal: calculated creatinine clearance (CrCl) ≥ 45 ml/min based on the original weight based Cockcroft and Gault formula
12. For women: Must be surgically sterile, postmenopausal, or compliant with a highly reliable contraceptive method (failure rate <1%) during and for 6 months after the treatment period; must have a negative serum or urine pregnancy test within 7 days before study enrollment and must not be breast-feeding.
13. For men: Must during chemotherapy take adequate contraceptive measures.

Exclusion Criteria:

1. Prior radiotherapy to the thorax.
2. Clinical superior vena cava syndrome, malignant pleural effusion or malignant pericardial effusion.
3. T4, specified as:Tumor growth in large blood vessels on spiral CT scan or encasement >50%
4. multiple nodules in the same or ipsilateral lobe(s).
5. Post-obstructive atelectasis or infiltration that cannot be distinguished from tumor on a CT-PET scan.
6. Patients with a diagnosis of other cancer within the last 3-years (except in situ carcinoma's and / or non-melanoma skin cancer).
7. Pregnant women, lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-05; Primary Completion 2020-12 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Local progression-free survival at 1 year | 1 year

SECONDARY OUTCOMES:
Toxicity | 1 year
Overall survival | 1 year
Quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: José Belderbos, MD, PhD, Principal Investigator — NKI-AvL
Locations (7):
- University Hospital Leuven, campus Gasthuisberg, Leuven, Belgium
- Rigshospitalet, Copenhagen, Denmark
- Netherlands (3):
  - MAASTRO clinic, Maastricht, Limburg
  - NKI/AVL, Amsterdam
  - Academic Medical Centre, Amsterdam
- Karolinska Hospital, Stockholm, Sweden
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooke SA, Belderbos JSA, Stam B, Reymen B, Lambrecht M, Fredberg Persson G, Faivre-Finn C, Dieleman EMT, van Diessen J, de Ruysscher D, Sonke JJ. Esophageal Toxicity After Dose-Escalated Radiation Therapy for Stage II-III Non-Small Cell Lung Cancer: A Secondary Analysis of the Phase 2 Randomized ARTFORCE PET-Boost Trial. Int J Radiat Oncol Biol Phys. 2025 Aug 1;122(5):1227-1237. doi: 10.1016/j.ijrobp.2025.03.001. Epub 2025 Mar 28. PMID 40156600
- [Derived] Cooke SA, de Ruysscher D, Reymen B, Lambrecht M, Fredberg Persson G, Faivre-Finn C, Dieleman EMT, Lewensohn R, van Diessen JNA, Sikorska K, Lalezari F, Vogel W, van Elmpt W, Damen EMF, Sonke JJ, Belderbos JSA. 18F-FDG-PET guided vs whole tumour radiotherapy dose escalation in patients with locally advanced non-small cell lung cancer (PET-Boost): Results from a randomised clinical trial. Radiother Oncol. 2023 Apr;181:109492. doi: 10.1016/j.radonc.2023.109492. Epub 2023 Jan 24. PMID 36706958
- [Derived] van Diessen J, De Ruysscher D, Sonke JJ, Damen E, Sikorska K, Reymen B, van Elmpt W, Westman G, Fredberg Persson G, Dieleman E, Bjorkestrand H, Faivre-Finn C, Belderbos J. The acute and late toxicity results of a randomized phase II dose-escalation trial in non-small cell lung cancer (PET-boost trial). Radiother Oncol. 2019 Feb;131:166-173. doi: 10.1016/j.radonc.2018.09.019. Epub 2018 Oct 13. PMID 30327236
- [Derived] Defraene G, La Fontaine M, van Kranen S, Reymen B, Belderbos J, Sonke JJ, De Ruysscher D. Radiation-Induced Lung Density Changes on CT Scan for NSCLC: No Impact of Dose-Escalation Level or Volume. Int J Radiat Oncol Biol Phys. 2018 Nov 1;102(3):642-650. doi: 10.1016/j.ijrobp.2018.06.038. Epub 2018 Jul 2. PMID 30244882
- [Derived] van Elmpt W, Zegers CML, Reymen B, Even AJG, Dingemans AC, Oellers M, Wildberger JE, Mottaghy FM, Das M, Troost EGC, Lambin P. Multiparametric imaging of patient and tumour heterogeneity in non-small-cell lung cancer: quantification of tumour hypoxia, metabolism and perfusion. Eur J Nucl Med Mol Imaging. 2016 Feb;43(2):240-248. doi: 10.1007/s00259-015-3169-4. Epub 2015 Sep 4. PMID 26338178